CLINICAL TRIAL: NCT06847451
Title: Red Cell Distribution Width as a Prognostic Factor for Morbidity and Mortality of Intensive Care Unit Patients With Sepsis.
Brief Title: Assessment of Red Cell Distribution Width's Prognostic Ability in Septic Intensive Care Unit Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MS85/2024
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-02

CONDITIONS: Sepsis
Keywords: sepsis; intensive care units; Red Cell Distribution Width; inflammatory markers; prognosis
MeSH Terms: conditions — Sepsis | interventions — Erythrocyte Indices

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — Whole blood samples, urine samples, sputum samples, skin swabs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Prognostic biomarker as Red Cell Distribution Width — Assessment of prognostic value of Red Cell Distribution Width in septic intensive care unit patients for 28 days mortality.
  Other Names: C-reactive proteins; Total leukocytic count; Serum lactate; Sequential Organ Failure Assessment (SOFA) Score

SUMMARY:
Various biomarkers are used for predicting outcome from sepsis and septic shock, but single value doesn't give a clear-cut picture. This prospective observational study aims to approach the prognostic value of Red Cell Distribution Width for morbidity and mortality of intensive care unit patients with sepsis. and this will be achieved by:

* Assessment of prognostic value of red cell distribution width in septic intensive care unit patients for 28 days mortality
* Comparison between red cell distribution width and other inflammatory markers as C-reactive protein and serum lactate as well as other scoring systems such as Sequential Organ Failure Assessment (SOFA) score, regarding their prognostic discriminative ability.

DETAILED DESCRIPTION:
Critically ill patients admitted to Ain Shams University hospital intensive care units who fulfill the criteria of sepsis and septic shock according to the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) will be enrolled.

All patients will be resuscitated and managed according to Ain Shams University Hospitals protocol for sepsis and septic shock.

On admission, and after applying the exclusion and inclusion criteria, all clinical data will be collected from participants, which will mainly include patient's detailed medical history, site of infection, blood routine test, biochemical test, other inflammatory markers as C-reactive protein, Arterial blood gas for serum lactate count, and cultures samples according to source of infection. Red cell distribution width will be recorded for each patient on admission, then patients will be followed up for 28 days mortality.

Patient's morbidity will be defined by Sequential Organ Failure Assessment (SOFA) Score, it will be calculated and recorded on admission and will be followed up as well.

ELIGIBILITY:
Inclusion Criteria:

* Age Group: all adult patients aged more than 18 Years old and less than 70 years old.
* Intensive care unit admitted patients with sepsis.

Exclusion Criteria:

* Patients less than 18 years old and more than 70 years old.
* Patients with known hematological disease (e.g., leukemia, myelodysplastic syndrome), human immunodeficiency virus (HIV) infection or any immunosuppressant usage history.
* Patients having uncured malignancy.
* Patients who had a cardiac arrest event before ICU arrival.
* Patients who had recent (less than one week) blood transfusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to Ain Shams University hospital intensive care units who fulfill the criteria of sepsis and septic shock according to the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
Assessment of prognostic value of Red Cell Distribution Width in septic Intensive care units patients for 28 days mortality. | 28 days
  Septic patients will be followed up at intensive care unit for a maximum duration of 28 days, patients will be divided then to survival and mortality groups and initial Red Cell Distribution Width value taken on admission will be reported for each individual to check relation between initial Red Cell Distribution Width reading and patients mortality. additionally, identifying a Red Cell Distribution Width cut-off value for both groups.

SECONDARY OUTCOMES:
Comparison between Red Cell Distribution Width and other inflammatory markers as well as known scoring systems regarding their prognostic discriminative ability. | 28 days
  Comparison between Red Cell Distribution and other inflammatory markers as C-reactive protein, Total leukocytic count, serum lactate as well as known scoring systems such as sequential organ failure assessment (SOFA) score regarding their prognostic discriminative ability for 28 days mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Farah H Barsoum, M.B.B.CH, Principal Investigator — Anesthesia resident Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be shared once study is completed
Supporting Information: Study Protocol, SAP
Access Criteria: free